CLINICAL TRIAL: NCT01765075
Title: Signal Transfer of Atrial Fibrillation Data to Guide Human Treatment
Acronym: STARLIGHT
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: STARLIGHT - 1012
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Permanent Atrial Fibrillation
Keywords: Electrophysiological mapping; Multi-electrode catheter

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing cardiac ablation for permanent AF

SUMMARY:
The purpose of the study is to gather electrophysiological data using a multi-electrode mapping catheter during a clinically indicated cardiac ablation procedure for the treatment of persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above, or above legal age and willing and capable of giving informed consent specific to national law
* Scheduled for a clinically indicated cardiac ablation for the treatment of persistent atrial fibrillation
* Able to meet study requirements for follow-up visit

Exclusion Criteria:

* Permanent leads or presence of prosthetic or severely stenotic tricuspid or mitral valves
* Active systemic infection or sepsis
* Echocardiographically confirmed presence of thrombus
* Atrial thrombus, myxoma, inter-atrial baffle patch or occluder device for those subjects in whom a transseptal approach is required
* Subjects who cannot be anticoagulated or infused with heparinized saline
* Heparin induced thrombocytopenia
* Hemodynamic instability or shock
* Atrial anatomy contradictory to catheter labeling or size indices
* EF < 35%
* Subjects with an active heart failure decompensation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Permanent atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Record 20 sets of electrophysiological data with a multi-electrode mapping catheter. | Acute - time of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jas Gill, MA MD FRCP FACC, Principal Investigator — Guys & St. Thomas' Hospital
Locations (2):
- Na Homolce, Prague, Czechia
- Guys & St. Thomas' Hospital, London, United Kingdom

REFERENCES:
- [Derived] Child N, Clayton RH, Roney CH, Laughner JI, Shuros A, Neuzil P, Petru J, Jackson T, Porter B, Bostock J, Niederer SA, Razavi RS, Rinaldi CA, Taggart P, Wright MJ, Gill J. Unraveling the Underlying Arrhythmia Mechanism in Persistent Atrial Fibrillation: Results From the STARLIGHT Study. Circ Arrhythm Electrophysiol. 2018 Jun;11(6):e005897. doi: 10.1161/CIRCEP.117.005897. PMID 29858382